CLINICAL TRIAL: NCT03698929
Title: A Randomized, Double-blind, Crossover Study on the Effect of Dietary Cholesterol on Plasma Lipids in Individuals With No Baseline Cholesterol Intake
Brief Title: Effect of Dietary Cholesterol on Plasma Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: PhysiciansCRM
Record Dates: First submitted 2018-09-25; First posted 2018-10-09 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Dietary Modification; Nutritional and Metabolic Disease
Keywords: dietary cholesterol; cholesterol; nutrition; egg yolks; eggs
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, crossover
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Effect of Cholesterol - Egg Phase (Active Comparator): In a randomized, 9-week crossover trial, we will test the effects of dietary cholesterol in individuals without baseline cholesterol intake through two 4-week dietary intervention periods, using baked goods containing egg yolks or egg-free baked goods. During the egg phase participants will consume two egg yolks a day for four weeks. Each week, participants will be given a week's worth of baked goods containing two egg yolks each.
  Interventions: Other: Dietary Effect of Cholesterol - Egg Phase
- Dietary Effect of Cholesterol - No-Egg Phase (Placebo Comparator): In a randomized, 9-week crossover trial, we will test the effects of dietary cholesterol in individuals without baseline cholesterol intake through two 4-week dietary intervention periods, using baked goods containing egg yolks or egg-free baked goods. During the no-egg phase participants will consume an egg-free product for four weeks. Each week participants will be given a week's worth of egg-free baked goods.
  Interventions: Other: Dietary Effect of Cholesterol - Non-Egg Phase

INTERVENTIONS:
Other: Dietary Effect of Cholesterol - Egg Phase — After the study entry, you will be assigned by chance, like the flip of a coin, to one of two groups. You will have an equal chance of being assigned to either group. Each group will be asked to consume baked goods daily. The two groups will consume the same baked goods, but in a different order. Each week, you will be given a week's worth of baked goods.
  Arms: Dietary Effect of Cholesterol - Egg Phase
Other: Dietary Effect of Cholesterol - Non-Egg Phase — After the study entry, you will be assigned by chance, like the flip of a coin, to one of two groups. You will have an equal chance of being assigned to either group. Each group will be asked to consume baked goods daily. The two groups will consume the same baked goods, but in a different order. Each week, you will be given a week's worth of baked goods.
  Arms: Dietary Effect of Cholesterol - No-Egg Phase

SUMMARY:
The Physicians Committee is carrying out a research study to improve the investigator's understanding and expand the literature to quantify the effect of foods on blood cholesterol. This study will measure changes in low density lipoprotein (LDL) concentration, sometimes called "bad cholesterol," over 2 study periods of 4 weeks each, with 1 rest week in between. Approximately 50 subjects will participate in this study.

DETAILED DESCRIPTION:
In a 9-week double-blind, crossover trial, participants will consume baked goods with either 2 egg yolks or an isocaloric egg-free product daily for 4 weeks. After a one-week washout period, participants will cross to the other dietary intervention. Participants will be asked not to make changes to their exercise patterns or diet, apart from consuming the provided products, for the study period. Changes in LDL cholesterol concentrations will be the primary dependent variable.

Study evaluations, known as health assessments, will be held at the Physicians Committee's office.

Group assignment: After the study entry, will be assigned by chance, like the flip of a coin, to one of two groups. The participant will have an equal chance of being assigned to either group. Each group will be asked to consume baked goods daily. The two groups will consume the same baked goods, but in a different order. The baked goods will be made from wheat flour with a small amount of sugar, salt, yeast, and other ingredients that are common to baked goods. There will be no animal-derived ingredients, except that some products will contain egg. Each week, the participant will be given a week's worth of baked goods.

ELIGIBILITY:
Inclusion Criteria:

• Following vegan diet for 6 or more months

Exclusion Criteria:

* Following vegan for less than 6 months
* Smoking during the past six months
* Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
* Pregnancy or intention to become pregnant during the study period
* Unstable medical or psychiatric illness
* Lack of English fluency
* Inability or unwillingness to participate in all components of the study
* Egg allergy
* Use of cholesterol-lowering medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Effect of Dietary Cholesterol on Plasma Lipids | 9 weeks total
  Examining the change of plasma lipids after consuming dietary cholesterol daily for one of two 4 week intervention periods with a 1 week washout period.

CONTACTS AND LOCATIONS:
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided